CLINICAL TRIAL: NCT03961464
Title: The Effect of NMDA Receptor Partial Agonist D-cycloserine on Emotional Processing, Stress and Memory in Healthy Volunteers
Brief Title: The Effect of D-cycloserine on Emotional Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R57491/RE001
Record Dates: First submitted 2019-03-04; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2018-06

CONDITIONS: Cycloserine; Healthy Volunteer
Keywords: Emotion processing; Autobiographical memory; Stress
MeSH Terms: interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- d-cycloserine (Experimental): oral, capsule, 250 mg
  Interventions: Drug: d-cycloserine
- Placebo (Experimental): oral, capsule, lactose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: d-cycloserine — Single dose
  Arms: d-cycloserine
Drug: Placebo — Single dose
  Arms: Placebo

SUMMARY:
To investigate the effects of N-methyl-D-aspartate (NMDA) partial agonist DCS on emotional processing, memory and stress tasks

DETAILED DESCRIPTION:
The aim of the present study is to assess the effect of DCS on emotional processing relevant to antidepressant drug activity. For this, 40 healthy volunteers will be recruited to the study and randomized to receive a single session of 250mg DCS or placebo. 3 hours and 24 hours after active drug/placebo administration, the effects of emotional processing via the use of cognitive tasks will be assessed. Also, given the important role of DCS in memory and stress, we also include tasks to explore changes in autobiographical memory and in psychological and physiological measures of stress and arousal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Willing and able to give informed consent for participation in the study
* Body mass index (BMI) within the range of 19-30kg/m2
* Sufficiently fluent English to understand and complete the task

Exclusion Criteria:

* Currently take any psychoactive medication.
* Have taken any CNS-active medication during the last 6 weeks.
* Currently take any medication with cycloserine, ethionamide or isoniazid
* Have suffered from any past or current psychiatric disorder (e.g. depression, anxiety)
* Have lifetime history of epilepsy or other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Have history of heart disease, significant hypertension
* Have history of Megaloblastic Anaemia, Sideroblastic Anaemia
* Have history of kidney disease with reduction in kidney function
* Have severe renal impairment
* Have suffered from lactose intolerance
* Are currently pregnant, breastfeeding or trying to get pregnant
* Have a current or past history of drug or alcohol dependency
* Have participated in a psychological or medical study involving the use of medication within the last 3 months
* Have previously participated in a study using the same, or similar, emotional processing tasks
* Smoke more than 5 cigarettes per day
* Have dyslexia (given the nature of the computer tasks)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Performance in a facial expression recognition task | 3 hours after drug/placebo administration
  Participants are presented with individual pictures of facial expressions of emotions. Each presented face displays one of six basic emotions (anger, disgust, fear, happiness, sadness, or surprise). Each emotional expression is presented at different levels of intensity which have been created by combining shape and texture features of the two extremes "neutral" (0%) and "full prototypical emotion" (100%) to varying degrees. Examples of neutral facial expressions are presented as well. Participants are instructed to correctly classify each facial expression as angry, disgusted, fearful, happy, sad, surprised or neutral both as quickly and as accurately as possible. Responses are made by pushing one out of seven labelled keys on a response box. Hit rates, false alarm rates, and reaction times for correct classifications are measured separately for each emotion.
Performance in an emotional recall task | 3 hours after drug/placebo administration
  Following a delay period after the emotional categorisation task (about 15 min), emotional recall memory is assessed. Participants are asked to recall and write down as many words as possible from the emotional categorization task. Numbers of correctly and incorrectly recalled positive and negative words are measured.
Performance in an autobiographical memory task | 3 hours after drug/placebo administration
  The autobiographical memory cues are presented visually on computer screen in a fixed order, with positive, negative, and neutral words alternating, each word will be presented only once. Participants are instructed that, for each cue word, they should respond with a memory of an autobiographical event which had lasted less than 1 day and which had occurred at a specific time and place. They are told that the event could have occurred recently or a long time ago and could have been important or trivial but that no responses should be repeated for a subsequent word. Correct and incorrect examples are given. Responses are tape-recorded for subsequent coding.

SECONDARY OUTCOMES:
Performance in an emotional categorisation task | 3 hours after drug/placebo administration
  Participants are presented with positive and negative personality descriptors and are asked to classify the valence of each word. These words describe either extremely agreeable/positive characteristics (e.g. "cheerful", "honest", "optimistic") or extremely disagreeable/negative characteristics (e.g. "domineering", "untidy", "hostile") and are presented individually in the centre of the screen. Participants are instructed to imagine themselves overhearing someone describing them with each of the words and to indicate as quickly and accurately as possible whether they would like or dislike to be described with each of the words. Responses are made by pressing a correspondingly labelled key on a button box. Reaction times for correct classifications are measured separately for positive and negative words.
Performance in an emotional faces dot probe task | 3 hours after drug/placebo administration
  Pictures of positive and negative emotional stimuli (happy and fearful facial expressions) are presented individually together with a matched neutral stimulus (neutral face). On each trial, one stimulus is shown above and the other below a central fixation point. Subsequently, a probe appears behind one of the stimuli and participants have to correctly classify the probe as quickly and as accurately as possible. Stimuli can be masked (i.e. presented very briefly and followed by a jumbled face) or unmasked (i.e. presented for a longer period without a subsequent masking stimulus). Reaction times for correct responses are recorded and vigilance scores are calculated for masked and unmasked positive and negative stimuli by subtracting reaction time data from trials when the probe appeared in the same position as the emotional stimulus (congruent trials) from trials when the probe appeared in the opposite position to the emotional stimulus (incongruent trials).
Performance in an emotional recognition task | Emotional recognition memory is assessed by presenting participants with the original personality descriptors plus an equal number of matched distractor words (50% positive, 50% negative). Participants are asked to ind
  3 hours after drug/placebo administration
Performance in a cognitive stress task | 3 hours after drug/placebo administration
  The computer stress task is designed to induce psychological stress.It is presented as a series of mental arithmetic, verbal and visuospatial challenges on the screen which participants are required to solve. In the stress condition, there is a time limit for completing each challenge, which is displayed on the screen as a time bar. To induce a high failure rate, the timing for each challenge is set depending on individual's previous performance at 10% less than the time that it took to previously correctly solve challenges. The difficulty of the challenges is automatically varied to ensure that participants are getting only 20-40% of the challenges correctly completed within the time. To ensure a high failure rate, some of the verbal challenges (anagrams) are impossible to solve. Participants are given feedback on their performance on the screen which indicates that they are performing badly.
Performance in a facial expression recognition task | 24 hours after drug/placebo administration
  Participants are presented with individual pictures of facial expressions of emotions. Each presented face displays one of six basic emotions (anger, disgust, fear, happiness, sadness, or surprise). Each emotional expression is presented at different levels of intensity which have been created by combining shape and texture features of the two extremes "neutral" (0%) and "full prototypical emotion" (100%) to varying degrees. Examples of neutral facial expressions are presented as well. Participants are instructed to correctly classify each facial expression as angry, disgusted, fearful, happy, sad, surprised or neutral both as quickly and as accurately as possible. Responses are made by pushing one out of seven labelled keys on a response box. Hit rates, false alarm rates, and reaction times for correct classifications are measured separately for each emotion.
Performance in an emotional recall task | 24 hours after drug/placebo administration
  Participants are asked to recall and write down as many words as possible from yesterday's emotional categorization task. Numbers of correctly and incorrectly recalled positive and negative words are measured.
Performance in an autobiographical memory task | 24 hours after drug/placebo administration
  The autobiographical memory cues are presented visually on computer screen in a fixed order, with positive, negative, and neutral words alternating, each word will be presented only once. Participants are instructed that, for each cue word, they should respond with a memory of an autobiographical event which had lasted less than 1 day and which had occurred at a specific time and place. They are told that the event could have occurred recently or a long time ago and could have been important or trivial but that no responses should be repeated for a subsequent word. Correct and incorrect examples are given. Responses are tape-recorded for subsequent coding.

OTHER OUTCOMES:
Change in subjective mood | 3 hours after drug/placebo administration
  Positive and Negative Affect Schedule. Standard questionnaire for subjectively felt positive and negative affect. Two scores: (1) Positive score: ranging from 10 to 50 (higher score representing greater extent of positive affect). (2) Negative score: ranging from 10 to 50 (higher score representing greater extent of negative affect).
Change in subjective anxiety | 3 hours after drug/placebo administration
  State Anxiety Inventory. Standard questionnaire for subjectively felt anxiety. State anxiety: ranging from 20 to 80 (higher scores indicating higher state anxiety levels).
Change in subjective energy | 3 hours after drug/placebo administration
  Zersen's Befindlichkeits-Skala. Standard questionnaire for subjectively felt mood and energy levels. Total score ranging from 0 to 112. Subscores: Mood (ranging from 0 to 94) and Energy (ranging from 0 to 18). Sum of subscores for mood and energy provide total score. Higher scores represent worse subjective mood and energy
Change in subjective state | 3 hours after drug/placebo administration
  Visual Analogue Scales of different subjective states (happy, sad, interested, anxious, stressed, hostile, nausea, dizziness, dry mouth, headache, alert, agitation). Minimum = 0 mm ("Not at all") , Maximum = 100 mm ("Extremely"). Greater scores represent greater extent of felt emotions/side effects.
Change in subjective anxiety for cognitive stress task | After cognitive stress task
  State Anxiety Inventory. Standard questionnaire for subjectively felt anxiety. State anxiety: ranging from 20 to 80 (higher scores indicating higher state anxiety levels).
Change in subjective mood for cognitive stress task | After cognitive stress task
  Positive and Negative Affect Schedule. Standard questionnaire for subjectively felt positive and negative affect. Two scores: (1) Positive score: ranging from 10 to 50 (higher score representing greater extent of positive affect). (2) Negative score: ranging from 10 to 50 (higher score representing greater extent of negative affect).
Change in subjective state for cognitive stress task | After cognitive stress task
  Visual Analogue Scales of different subjective states (happy, sad, interested, anxious, stressed, hostile, nausea, dizziness, dry mouth, headache, alert, agitation). Minimum = 0 mm ("Not at all") , Maximum = 100 mm ("Extremely"). Greater scores represent greater extent of felt emotions/side effects.
Physiological measures (Skin Conductance Response) for cognitive stress task | During cognitive stress task
  The skin conductance response (SCR), also known as the electrodermal response is the phenomenon that the skin momentarily becomes a better conductor of electricity when either external or internal stimuli
Physiological measures (blood pressure) for cognitive stress task | During cognitive stress task
  Systolic and diastolic blood pressure are the two values that determine whether participant's blood pressure is normal, too high or too low.
Change in subjective mood | 24 hours after drug/placebo administration
  Positive and Negative Affect Schedule. Standard questionnaire for subjectively felt positive and negative affect. Two scores: (1) Positive score: ranging from 10 to 50 (higher score representing greater extent of positive affect). (2) Negative score: ranging from 10 to 50 (higher score representing greater extent of negative affect).
Change in subjective anxiety | 24 hours after drug/placebo administration
  State Anxiety Inventory. Standard questionnaire for subjectively felt anxiety. State anxiety: ranging from 20 to 80 (higher scores indicating higher state anxiety levels).
Change in subjective energy | 24 hours after drug/placebo administration
  Zersen's Befindlichkeits-Skala. Standard questionnaire for subjectively felt mood and energy levels. Total score ranging from 0 to 112. Subscores: Mood (ranging from 0 to 94) and Energy (ranging from 0 to 18). Sum of subscores for mood and energy provide total score. Higher scores represent worse subjective mood and energy
Change in subjective state | 24 hours after drug/placebo administration
  Visual Analogue Scales of different subjective states (happy, sad, interested, anxious, stressed, hostile, nausea, dizziness, dry mouth, headache, alert, agitation). Minimum = 0 mm ("Not at all") , Maximum = 100 mm ("Extremely"). Greater scores represent greater extent of felt emotions/side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided